CLINICAL TRIAL: NCT04476446
Title: An Open-Label Expanded Access Protocol for Esketamine Treatment of Subjects With Treatment Resistant Depression (TRD) Who do Not Have Other Treatment Alternatives
Brief Title: An Expanded Access Protocol for Esketamine Treatment in Participants With Treatment Resistant Depression (TRD) Who do Not Have Other Treatment Alternatives
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108690; 54135419TRD4006 (Other: Janssen-Cilag, S.A.)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intranasal Esketamine (Experimental): Induction Phase: Participants will self-administer esketamine intranasally 56 milligram (mg) on Day 1 followed by 56 mg or 84 mg (as a flexible dose regimen) twice per week for 4 weeks. Participants greater than or equal to (>=) 65 years old will start at a dose of 28 mg on Day 1. Maintenance Phase: Participants will self-administer esketamine 56 mg or 84 mg intranasally once per week from Week 5 to Week 9. Subsequently from Week 9, based on the investigator's clinical judgment, participants will self-administer esketamine 56 mg or 84 mg intranasally once or twice a week.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Participants will receive esketamine at doses of either 56 mg or 84 mg intranasally once or twice a week based on the investigator's clinical judgment.
  Other Names: JNJ-54135419

SUMMARY:
The purpose of this expanded access program (EAP) is to provide expanded access to esketamine treatment and collect additional safety data and quality of life until esketamine is commercially available for participants with Treatment-Resistant Depression (TRD).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have an unmet medical need to treat treatment-resistant depression (TRD) with Esketamine Nasal Spray, an investigational compound, that has not been approved the local health authority. This means no other treatment options are available and the participant must be unable to participate in a clinical trial; for example, because they do not fulfill the eligibility criteria of the protocol or there are no trial sites within a reasonable distance of where they reside
* Participant must not participate in a clinical trial or be concurrently treated with an investigational drug when being treated with Esketamine Nasal Spray
* Participants must have TRD with the diagnosis verified by a psychiatrist, and have exhausted all other options including all alternative treatment options with marketed therapies, specifically (a) Participants must meet the Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM)-5 diagnostic criteria for single-episode major depressive episode (MDD) (if single-episode MDD, the duration must be 2 years) or recurrent MDD, without psychotic features (b) Participants must have had nonresponse to 2 or more oral antidepressant (of the same or a different class) treatments in the current episode of depression confirmed by documented medical history and/or pharmacy/prescription records i.e., treatments were prescribed in adequate dosages for adequate duration with affirmation of treatment adherence, to meet criteria for TRD, and have failed at least one augmentation/combination strategy and have failed an adequate course (greater than or equal to [>=] 7 sessions) of, or have a contraindication/no access or refuses electro-convulsive therapy (ECT)
* Participants must have exhausted clinical trials, early access programs or named patient programs that may be available in your region
* Participants must have moderate to severe depression per clinical judgement
* Participants must be medically stable based on physical examination, medical history, vital signs (including stable blood pressure) and 12-lead electrocardiogram (ECG) performed prior to dosing
* Participants must be medically stable based on clinical laboratory tests (complete blood count (CBC), chemistry, liver enzymes and thyroid stimulating hormone [TSH]) performed prior to first dose
* Participants must be comfortable with self-administration of intranasal medication and be able to follow the intranasal administration instructions provided
* Before the start of dosing, a woman must be either: non-childbirth potential or practicing a highly effective method of birth control consistent with local regulations. Men must agree to use a barrier method of birth control.
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) before dosing begins and a negative urine pregnancy test each time tested
* Participants must be willing and able to adhere to the prohibitions and restrictions specified for study
* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for early access program (EPA) and is willing to participate in the EPA, if required by law or regulation

Exclusion Criteria:

* The participant's depressive symptoms have previously demonstrated nonresponse to Esketamine Nasal Spray or ketamine in the current major depressive episode per clinical judgment
* Participant has a current or prior Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnosis of a psychotic disorder or major depressive episode (MDD) with psychosis, bipolar or related disorders, or intellectual disability (only DSM-5 diagnostic code 319).
* Participant has homicidal ideation/intent or has suicidal ideation with some intent to act within 6 months per the requesting psychiatrist's clinical judgment
* Participant has a history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria, except nicotine or caffeine, within 6 months before the start of the first dose. (a). A history (lifetime) of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3, 4-methylenedioxy-methamphetamine (MDMA) hallucinogen-related use disorder is exclusionary
* Participants with active seizures (uncomplicated childhood febrile seizures with no sequelae are not exclusionary). Participants with a history of seizure are allowed provided that seizures are controlled, and no seizure has been experienced in the 6 months prior to expanded access protocol (EAP) entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 6 months
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Change from Baseline in European Quality of Life (EuroQol) Group, 5-Dimension, 5-Level (EQ 5D-5L) | Up to 6 months
  The EQ-5D-5L is a standardized instrument used as a measure of health outcome, designed for self-completion by respondents. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems. Where Level 1: no problem, Level 2: slight problems, Level 3: moderate problems, Level 4: severe problems and Level 5: extreme problems).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag, S.A. Clinical Trial, Study Director — Janssen-Cilag, S.A.
Locations (8):
- Mexico (8):
  - Clínica de Ansiedad, Depresión y Estrés CADE, S. de R.L. de C.V., Guadalajara
  - Gabipros SC., Mexico City
  - Avalon Vinculación Médica En Salud Mental, Mexico City
  - Hospital Espanol, Mexico City
  - Ketamine Mexico S. de RL. de C.V., Mexico City
  - Ángel Alberto Ruiz Chow, México
  - Especialidades en Neuropsiquiatría de México S.C., México
  - Clínica de Interdisciplinas Congnitivo Conductuales, México

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency